CLINICAL TRIAL: NCT04499508
Title: APPLY Study: A Prospective, Single Center Study Appraising the Embolization of Aneurysms Using the Balt Optima™ Coil System
Brief Title: Appraising the Embolization of Aneurysms Using Balt Optima™ Coil System (APPLY Study)
Acronym: APPLY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vascular Neurology of Southern California Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VNSC-022020
Record Dates: First submitted 2020-07-28; First posted 2020-08-05 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Aneurysm; Intracranial Aneurysm; Ruptured Aneurysm; Subarachnoid Hemorrhage, Aneurysmal; Cerebral Aneurysm Unruptured
Keywords: Brain aneurysm; Optima Coil System; Endovascular Coiling; Embolization; Ruptured Intracranial Aneurysm; Unruptured Intracranial Aneurysm
MeSH Terms: conditions — Aneurysm; Intracranial Aneurysm; Aneurysm, Ruptured; Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, single-center, post-market, real-world, investigator-initiated study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment with Optima Balt Coils (Experimental): The APPLY study is a single-arm prospective study which means that everyone enrolled in the clinical trial will be/has been treated with the Optima Balt Coils.
  Interventions: Device: Optima Coil System

INTERVENTIONS:
Device: Optima Coil System — Patients who have qualified for endovascular coiling in effort to treat intracranial aneurysms were treated with
  Other Names: Embolization of Intracranial Aneurysm; Optima Balt Coil System; Neurovascular Embolization Device

SUMMARY:
In recent years, many developments have been made to the tools and techniques used to treat IAs via endovascular intervention. Specifically, to the detachable coils themselves. In March 2018, the US Food and Drug administration granted Balt USA 510(k) clearance for the Optima Coil System™. Earlier this year, the list of devices included within the system has expanded to include OptiMAX Complex Super Soft and Complex Soft coils. It consists of coils that come in Standard, Soft and Super Soft profiles and allows for instant detachment from the pusher. The APPLY study is a prospective, single-center investigator-initiated study meant to assess the use of the Balt Optima™ Coil System. The site is looking to enroll approximately 30 subjects over the course of two years. The Optima Coil System™ is commercially available in the United States as such this study is looking for real-world data.

DETAILED DESCRIPTION:
Intracranial aneurysms both ruptured and unruptured collectively affect a significant portion of the general population. Cases of unruptured intracranial aneurysms (UIA) are estimated to affect roughly 3% of the general population and aneurysmal subarachnoid hemorrhage (aSAH) has an incidence of 8 to 9 people per 100,000. There are two well-established treatment options for patients diagnosed with intracranial aneurysms (IA): surgical clipping and endovascular coiling. Neurosurgical intervention requires a craniotomy followed by the clipping of the aneurysm. Endovascular repair is minimally invasive as access to the afflicted vessel is gained through the femoral artery with the assistance of imaging guidance. During embolization, the aneurysm is occluded using coils of varying length, diameter, and softness. By filling the dome of the aneurysm physicians aim to prevent further blood flow into the bulge which will prevent the aneurysm from rupturing. In addition to coiling a stent may be placed to function as a blood flow diverting device.

The first-ever recorded use of coils in the treatment of intracranial aneurysms by way of endovascular intervention was in 1988. In 1989, detachable coils were designed by Guido Guglielmi, an endovascular neurosurgeon, who pioneered the concept of coil embolization. Since then, endovascular embolization has become effective, and in some cases preferred, method of treatment of intracranial aneurysms. A 2005 randomized, multicenter study titled International Subarachnoid Aneurysm Trial (ISAT) demonstrated that in comparison to surgical clipping, endovascular repair clinical outcomes result in significant risk reduction and long-term independence post-procedure. To verify their findings the ISAT authors reviewed the clinical outcomes at 1 year of 1063 of 1072 patients who underwent ruptured aneurysm embolization using detachable coils compared to 1055 of 1070 who were designated to neurosurgical clipping. At the one-year mark patients who experienced endovascular repair demonstrated poor prognosis with less frequency, as measured by mortality and extent of dependency, in 23.5% of cases in comparison to 30.9% of subjects treated via neurosurgical intervention. While the results seem to show a considerable preference for embolization, the patients in this designated sample were found to experience rebleeds at a higher frequency. Beyond resurgence of hemorrhaging, embolization risks include aneurysm perforation and/or rupture, thromboembolic events, and coil herniation out of the occluded site. Despite the aforementioned risk factors, it has become clear that embolization with detachable coils is a much safer treatment option as the rate of procedure-related complications is relatively low. This is true for patients with unruptured and ruptured intracranial aneurysms-size and location did not show any statistically significant impact.

The study will enroll approximately 30 subjects to allow us to adequately observe the benefits of the central limit theorem. Based on prior experience, we expect that approximately 10% of all participants may be lost to follow-up and/or will withdraw from the study. It is estimated that two years are needed to complete the study. The first year will be necessary to enroll 30 subjects and the second year will be necessary to complete the 12-month follow-up visits and study close out procedures. The device is to be used per Instructions for Use as indicated for treatment of intracranial aneurysms by way of coil embolization. Participating in this study will not contribute or be of detriment in any way of a subject's medical care. All study related data gathering activities are standard of care and do not require any special actions.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18
* Patients undergoing the embolization of large or small intracranial aneurysms
* Patient's physician has decided that the best treatment for the patient's neurovascular abnormalities is the Optima Coil System and the patient has agreed to the treatment
* Of the total number of coils implanted Optima™ Coil System accounts for at least 80%
* Fully executed IRB approved Informed Consent

Exclusion Criteria:

* Patient participation in another study that may disrupt the results of this study
* Anticipated life expectancy of less than 12-months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2023-04-09 (Estimated); Study Completion 2023-04-09 (Estimated)

PRIMARY OUTCOMES:
Occlusion Rates | 12 Months
  Successful occlusion rates defined as Raymond-Roy Occlusion Class I and II.
Mortality | 12 Months
  All-cause mortality.

SECONDARY OUTCOMES:
Occlusion Scale Score | Immediately post-procedure, 3-Months, and 12-Months
  Raymond-Roy Occlusion classification is measured via angiographic imaging of endovascularly treated intracranial aneurysms. The classes are the following: Class I indicates complete obliteration of the aneurysm. Class II indicates that post-coiling some residual neck is left. Class IIIa indicates residual aneurysm remains after coiling but these are likely to improve to Class I or II over time. Class IIIb indicates residual aneurysm remains but these are wider and larger, they also have a higher retreatment rate. Ideal aneurysm coiling classification post procedure is Class I, Class II, and in some cases Class IIIa.
Modified Rankin Scale (mRS) | Up to 1 year during various scheduled visits. Specifically, at discharge from hospital, at 3-month follow up and again at 12-months.
  Good Clinical Outcome defined as mRS = 0 - 2. The modified Rankin Scale measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other neurological disability via interview of subject or family. The scale ranges from 0 to 6, with 0 being the best outcome and 6 being the worst. Score 0 = patient shows no symptoms. Score 1 = no significant disability despite some symptoms, but patient is able to carry out all usual duties/activities. Score 2 = slight disability, patient is unable to carry out all previous activities but is able to look after their own affairs. Score 3 = moderate disability, requiring some help, but able to walk without assistance. Score 4 = moderate severe disability, patient is unable to walk and/or attend to their own bodily needs. Score 5 = severe disability, patient is bedridden, incontinent and requires constant nursing care. Score 6 = patient has expired.
Packing Density | Result is known immediately post-procedure.
  Number of coils necessary for packing density
Fluro Time | Result is known immediately post-procedure.
  Fluro time per case.
Other Devices Used | Result is known immediately post-procedure.
  Use of adjuncts, stent/balloon/Comaneci
Complications | At all time points from procedure to 12 Months.
  Major complications (i.e. intraoperative complications: inadvertent coil detachment, rupture/re-rupture, retreatment)
SAE | At all time points from procedure to 12 Months.
  Serious Adverse Events post-procedure at discharge, 3-months, and through the final 12-month visit-device related or otherwise.
Thromboembolic Events | At all time points from procedure to 12 Months.
  Post-treatment major thromboembolic events are defined as stroke events that occur immediately after the index procedure. Post endovascular coiling subjects are often at risk for stroke, this occurs as a formation in the blood vessel of a clot breaks loose and is carried by the blood stream and occludes another vessel. Thromboembolic events represent one of the most serious complications of embolization therapy, due to the possibility of permanent neurologic disability and death. As such these events will be closely monitored. This is not a quantitative or qualitative measurement but rather an archive of the circumstances should an event occur.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad A Taqi, MD, Principal Investigator — Vascular Neurology of Southern California; Anastasia Vechera, BA, Study Director — Vascular Neurology of Southern California
Locations (1):
- Vascular Neurology of Southern California, Thousand Oaks, California, United States

REFERENCES:
- [Background] Molyneux AJ, Kerr RS, Yu LM, Clarke M, Sneade M, Yarnold JA, Sandercock P; International Subarachnoid Aneurysm Trial (ISAT) Collaborative Group. International subarachnoid aneurysm trial (ISAT) of neurosurgical clipping versus endovascular coiling in 2143 patients with ruptured intracranial aneurysms: a randomised comparison of effects on survival, dependency, seizures, rebleeding, subgroups, and aneurysm occlusion. Lancet. 2005 Sep 3-9;366(9488):809-17. doi: 10.1016/S0140-6736(05)67214-5. PMID 16139655
- [Background] Yoo E, Kim DJ, Kim DI, Lee JW, Suh SH. Bailout stent deployment during coil embolization of intracranial aneurysms. AJNR Am J Neuroradiol. 2009 May;30(5):1028-34. doi: 10.3174/ajnr.A1482. Epub 2009 Feb 4. PMID 19193745
- [Background] Frazer D, Ahuja A, Watkins L, Cipolotti L. Coiling versus clipping for the treatment of aneurysmal subarachnoid hemorrhage: a longitudinal investigation into cognitive outcome. Neurosurgery. 2007 Mar;60(3):434-41; discussion 441-2. doi: 10.1227/01.NEU.0000255335.72662.25. PMID 17327787
- [Background] Jalbert JJ, Isaacs AJ, Kamel H, Sedrakyan A. Clipping and Coiling of Unruptured Intracranial Aneurysms Among Medicare Beneficiaries, 2000 to 2010. Stroke. 2015 Sep;46(9):2452-7. doi: 10.1161/STROKEAHA.115.009777. Epub 2015 Aug 6. PMID 26251248
- [Background] Guglielmi G. History of endovascular endosaccular occlusion of brain aneurysms: 1965-1990. Interv Neuroradiol. 2007 Sep;13(3):217-24. doi: 10.1177/159101990701300301. Epub 2007 Sep 15. PMID 20566113
- [Background] Katsaridis V, Papagiannaki C, Violaris C. Guglielmi detachable coils versus matrix coils: a comparison of the immediate posttreatment results of the embolization of 364 cerebral aneurysms in 307 patients: a single-center, single-surgeon experience. AJNR Am J Neuroradiol. 2006 Oct;27(9):1841-8. PMID 17032854
- [Background] Tamatani S, Ito Y, Abe H, Koike T, Takeuchi S, Tanaka R. Evaluation of the stability of aneurysms after embolization using detachable coils: correlation between stability of aneurysms and embolized volume of aneurysms. AJNR Am J Neuroradiol. 2002 May;23(5):762-7. PMID 12006273
- [Background] Ayling OG, Ibrahim GM, Drake B, Torner JC, Macdonald RL. Operative complications and differences in outcome after clipping and coiling of ruptured intracranial aneurysms. J Neurosurg. 2015 Sep;123(3):621-8. doi: 10.3171/2014.11.JNS141607. Epub 2015 Jun 5. PMID 26047409
- [Background] Mascitelli JR, Moyle H, Oermann EK, Polykarpou MF, Patel AA, Doshi AH, Gologorsky Y, Bederson JB, Patel AB. An update to the Raymond-Roy Occlusion Classification of intracranial aneurysms treated with coil embolization. J Neurointerv Surg. 2015 Jul;7(7):496-502. doi: 10.1136/neurintsurg-2014-011258. Epub 2014 Jun 4. PMID 24898735
- [Background] Hunt WE, Hess RM. Surgical risk as related to time of intervention in the repair of intracranial aneurysms. J Neurosurg. 1968 Jan;28(1):14-20. doi: 10.3171/jns.1968.28.1.0014. No abstract available. PMID 5635959
- [Background] van Swieten JC, Koudstaal PJ, Visser MC, Schouten HJ, van Gijn J. Interobserver agreement for the assessment of handicap in stroke patients. Stroke. 1988 May;19(5):604-7. doi: 10.1161/01.str.19.5.604. PMID 3363593
- [Result] Brilstra EH, Rinkel GJ, van der Graaf Y, van Rooij WJ, Algra A. Treatment of intracranial aneurysms by embolization with coils: a systematic review. Stroke. 1999 Feb;30(2):470-6. doi: 10.1161/01.str.30.2.470. PMID 9933290